CLINICAL TRIAL: NCT01868542
Title: A 20-week, Randomised, Multi-centre, Open-labelled Trial Comparing the Glycaemic Control of Levemir® Administered Once Daily According to Two Titration Algorithms (3-0-3 Algorithm and 2-4-6-8 Algorithm) After 20 Weeks in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin Treatment in Korea
Brief Title: A Trial Comparing the Glycaemic Control of Levemir® Administered Once Daily According to Two Insulin Detemir Titration Algorithms After 20 Weeks in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin Treatment With or Without Other Anti-diabetic Drugs (OADs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3994; U1111-1132-9267 (Other: WHO)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-0-3 Algorithm (Experimental): A once daily dosage of Insulin detemir (Levemir®) 100 U/mL 3 mL FlexPen® for subcutaneous administration was selected for this trial.During the treatment period insulin detemir was adjusted by the subject themselves (self-titration). Self-titration was performed every 3 days based on the lowest of three previous consecutive pre-breakfast SMPG values.Based on this glucose value, self-adjustment of insulin detemir dose was done. Metformin and Sulfonlylurea were allowed as OADs. For SMPG values, the following insulin detemir dose adjustments were done : >6.1 mmol/L (>110 mg/dL) +3U insulin detemir, 4.4-6.1 mmol/L (80-100 mg/dL) No adjustment in insulin detemir, < 4.4 mmol/L (<80 mg/dL) -3U insulin detemir.
  Interventions: Drug: insulin detemir
- 2-4-6-8 Algorithm (Experimental): A once daily dosage of Insulin detemir (Levemir®) 100 U/mL 3 mL FlexPen® for subcutaneous administration was selected for this trial. During the treatment period insulin detemir was adjusted by the subject themselves (self-titration). Self-titration was performed every 3 days based on the lowest of three previous consecutive pre-breakfast SMPG values.Based on this glucose value, self-adjustment of insulin detemir dose was done. Metformin and Sulfonlylurea were allowed as OADs. For SMPG values , the following insulin detemir dose adjustments were done : >10.0 mmol/L (180 mg/dL) +8U insulin detemir, 9.1-10.0 mmol/L (163-180 mg/dL) +6U insulin detemir, 8.1-9.0 mmol/L (145-162 mg/dL) +4 U insulin detemir, 7.1-8.0 mmol/L (127-144 mg/dL) +2U insulin detemir, 6.1-7.0 mmol/L (109-126 mg/dL) +2U insulin detemir, 4.1-6.0 mmol/L (73-108 mg/dL) No adjustment in insulin detemir, 3.1-4.0 mmol/L (56-72 mg/dL) -2U insulin detemir, <3.1 mmol/L (<56 mg/dL) -4U insulin detemir.
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Insulin detemir was administered once daily to the subjects. The dose was titrated based on the previous breakfast SMPG values.

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to compare the glycaemic control of Levemir® (insulin detemir) administered once daily according to two titration algorithms after 20 weeks in subjects with type 2 diabetes inadequately controlled on metformin treatment with or without other anti-diabetic drugs (OADs).

ELIGIBILITY:
Inclusion Criteria:

* - Diagnosed with type 2 diabetes mellitus at least 3 months prior to Visit 1 (week -2)
* - Treatment with at least 1000 mg metformin per day with/without other OADs at a stable dose (at either the maximal tolerated dose or at least half of the maximum recommended dose according to the package insert) for at least 3 months prior to Visit 1
* - Insulin-naïve subjects
* - HbA1c above or equal to 7.5% by central laboratory analysis
* - Body mass index (BMI) below or equal to 35.0 kg/m^2

Exclusion Criteria:

* - Female who is breast-feeding
* - The receipt of any investigational product within 4 weeks prior to Visit 1
* - Any contraindication to insulin detemir according to the domestic labelling
* - Anticipated change of dose of any systemic treatment with products, which in the investigator's opinion could interfere with glucose metabolism (such as systemic corticosteroids, beta-blockers, monoamine oxidase [MAO] inhibitors)
* - Clinically significant diseases which, in the investigator's opinion, may confound the results of the trial or pose additional risk in administering trial product
* - Any conditions that the investigator judges would interfere with trial participation or evaluation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Daejeon, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 6 sites in 1 country: South Korea
Groups:
- Insulin Detemir (3-0-3 Algorithm ): A once daily dosage of Insulin detemir (Levemir®) 100 U/mL 3 mL FlexPen® for subcutaneous administration was selected for this trial.During the treatment period insulin detemir was adjusted by the subject themselves (self-titration). Self-titration was performed every 3 days based on the lowest of three previous consecutive pre-breakfast SMPG values.Based on this glucose value, self-adjustment of insulin detemir dose was done. Metformin and Sulfonlylurea were allowed as OADs. For SMPG values , the following insulin detemir dose adjustments were done : >6.1 mmol/L (>110 mg/dL) +3U insulin detemir, 4.4-6.1 mmol/L (80-100 mg/dL) No adjustment in insulin detemir, < 4.4 mmol/L (<80 mg/dL) -3U insulin detemir.
- Insulin Detemir (2-4-6-8 Algorithm ): A once daily dosage of Insulin detemir (Levemir®) 100 U/mL 3 mL FlexPen® for subcutaneous administration was selected for this trial.During the treatment period insulin detemir was adjusted by the subject themselves (self-titration). Self-titration was performed every 3 days based on the lowest of three previous consecutive pre-breakfast SMPG values.Based on this glucose value, self-adjustment of insulin detemir dose was done. Metformin and Sulfonlylurea were allowed as OADs. For SMPG values , the following insulin detemir dose adjustments were done : >10.0 mmol/L (180 mg/dL) +8U insulin detemir, 9.1-10.0 mmol/L (163-180 mg/dL) +6U insulin detemir, 8.1-9.0 mmol/L (145-162 mg/dL) +4 U insulin detemir, 7.1-8.0 mmol/L (127-144 mg/dL) +2U insulin detemir, 6.1-7.0 mmol/L (109-126 mg/dL) +2U insulin detemir, 4.1-6.0 mmol/L (73-108 mg/dL) No adjustment in insulin detemir, 3.1-4.0 mmol/L (56-72 mg/dL) -2U insulin detemir, <3.1 mmol/L (<56 mg/dL) -4U insulin detemir.
Period: Overall Study
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Started | 23 | 23
Completed | 23 | 21
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Unclassified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm ) | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 6 | 4 | 10
Gender [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) From Baseline.
Description: Change in glycosylated haemoglobin A1c (HbA1c) (%) from baseline after 20 weeks of treatment. Only the subjects in the full analysis set with HbA1c values after 20 weeks of treatment were included.
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) - included all randomised subjects. 2 subjects withdrew after randomisation in the detemir (2-4-6-8 algorithm) arm.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 21
Percent (%) glycosylated haemoglobin | -0.9 (1.3) | -1.0 (1.2)

2. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c at 12 weeks of treatment from visit 2.
Time Frame: Week 0, week 12
Population: Full analysis set (FAS) - included all randomised subjects. 2 subjects withdrew after randomisation in the detemir (2-4-6-8)algorithm arm.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 21
Percent (%) glycosylated haemoglobin | -0.8 (1.3) | -0.9 (1.2)

3. Secondary Outcome: Proportion of Subjects Achieving HbA1c Below 7.0%
Description: Responder was a dichotomous endpoint (responder/non-responder) that was defined based on whether a subject had met the ADA HbA1c target at end of trial (HbA1c < 7.0% at end of trial) during 20 weeks of treatment.
Time Frame: Week 20
Population: Full analysis set (FAS) - included all randomised subjects. 2 subjects withdrew after randomisation in the detemir (2-4-6-8 algorithm ) arm.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 21
percentage (%) of subjects
  week 20 (Yes) | 8.7 | 14.3
  week 20 (No) | 91.3 | 85.7

4. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline
Description: Change in fasting plasma glucose from baseline.
Time Frame: week 0, week 12
Population: Full analysis set (FAS) - included all randomised subjects.2 subjects withdrew after randomisation in the detemir (2-4-6-8 algorithm) arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 21
mg/dL | -74.3 (73.0) | -44.6 (88.8)

5. Secondary Outcome: Incidence of Hypoglycaemic Episodes : Nocturnal (23:00-05:59) and Over 24 Hours.
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode occurred after the first administration of the investigational medicinal product (IMP), and no later than the last day on trial product. Hypoglycaemic episodes were defined as nocturnal if the time of onset was between 23:00 and 05:59 inclusive. All plasma glucose values: · equal or below 3.9 mmol/L (70 mg/dL) or · higher than 3.9 mmol/L (70 mg/dL) when they occur in conjunction with hypoglycaemic symptoms.
Time Frame: For 20 weeks of treatment and over 24 hours
Population: Safety Analysis Set (SAS): Included all subjects receiving at least one dose of trial product. Subjects contributed to the evaluation "as treated".
Measure: Number; unit: Episodes
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 23
Episodes
  Hypoglycaemic episodes | 72 | 119
  Nocturnal hypoglycaemic episodes | 22 | 17

6. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline
Description: Change in fasting plasma glucose from baseline.
Time Frame: Week 0, week 20
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 21
mg/dL | -60.4 (71.5) | -70.0 (63.8)

7. Secondary Outcome: Incidence of Adverse Events
Description: A treatment emergent adverse event (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than the day of visit 22.(week 20)
Time Frame: Week 20
Population: Safety analysis set - included all subjects receiving at least one dose of the trial product. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: events
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Number analyzed (Participants) | 23 | 23
events
  Treatment Emergent Adverse Events (TEAEs) | 24 | 29
  Serious Adverse Events (SAEs) | 0 | 1
  Non Serious Adverse Events (NSAEs) | 24 | 28

ADVERSE EVENTS:
Time Frame: A treatment emergent adverse event (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than the day of visit 22.
Description: Safety analysis set - included all subjects receiving at least one dose of the trial product. Subjects in the safety set contributed to the evaluation "as treated"
Arm/Group | Insulin Detemir (3-0-3 Algorithm ) | Insulin Detemir (2-4-6-8 Algorithm )
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/23
Other Adverse Events (participants affected / at risk) | 7/23 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (3-0-3 Algorithm ) (N=23) | Insulin Detemir (2-4-6-8 Algorithm ) (N=23)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (3-0-3 Algorithm ) (N=23) | Insulin Detemir (2-4-6-8 Algorithm ) (N=23)
Nasopharyngitis (Infections and infestations) | 3 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.